CLINICAL TRIAL: NCT02854579
Title: Safety and Efficacy Study of Neural Progenitor Cell Transplantation and Paracrine Factors From Human Mesenchymal Stem Cells to Treat Newborn With Hypoxic-ischemic Encephalopathy
Brief Title: Neural Progenitor Cell and Paracrine Factors to Treat Hypoxic Ischemic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Bethune International Peace Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Hunan Children's Hospital (Other Government); Shangluo Central Hospital (Other); 252 Military Hospital (Unknown)
Responsible Party: Principal Investigator, Zuo Luan, Principal Investigator, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NavyGHB-P-01
Record Dates: First submitted 2014-04-27; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Hypoxic-Ischemic Encephalopathy; progenitor cell; paracrine factor; adipose mesenchymal stem cell; neonate
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Neural progenitor cell (Experimental): Three doses of Neural progenitor cell (4*10^6) intrathecally at 48-72h, 5d and 10d after birth.+routine therapy
  Interventions: Biological: neural progenitor cell
- Paracrine factors (Experimental): Three doses of concentrated paracrine factors of human mesenchymal stem cell （0.5ml） intrathecally at 12h,24h,48h after birth.+routine therapy
  Interventions: Biological: Paracrine factors
- Progenitor cell and paracrine factors (Experimental): Three doses of concentrated paracrine factors 0.5ml intrathecally at 12h,24h,48h after birth.And three doses of neural progenitor cell (4*10^6) intrathecally at 48-72h, 5d and 10d after birth.+routine therapy
  Interventions: Biological: progenitor cell and paracrine factors
- Routine therapy (No Intervention): neonates only receive routine therapy

INTERVENTIONS:
Biological: neural progenitor cell — Neural progenitor cells are derived from the same aborted human fetal forebrain.
  Arms: Neural progenitor cell
Biological: Paracrine factors — The factors obtained from cultured human mesenchymal stem cells were concentrated 50 times
  Other Names: paracrine factor of human mesenchymal stem cells
  Arms: Paracrine factors
Biological: progenitor cell and paracrine factors — Neural progenitor cells will be received after paracrine factors therapy
  Arms: Progenitor cell and paracrine factors

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of allogenic neural progenitor cell and paracrine factors of human mesenchymal stem cells for patients with moderate/severe Hypoxic-Ischemic Encephalopathy

DETAILED DESCRIPTION:
Neonates diagnosed moderate/severe Hypoxic-Ischemic Encephalopathy after birth will receive routine therapy and be randomized to four arms for allogenic neural progenitor cells transplantation，paracrine factors of human mesenchymal stem cells intrathecal injection，combination of cell and factor or only routine therapy. Patients will be followed for neurodevelopmental outcome at 12 and 18 months in Pediatrics of Navy General Hospital. Magnetic Resonance Imaging, electroencephalogram, Bailey scores, Peabody development measure scale and Gross motor function measure assessment will be obtained in the following research.Results will be analyzed and described in study reports.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age ≥ 34weeks, body weight ≥ 2kg.
2. 1 minute apgar score ≤3, and 5 minutes apgar score ≤5, OR umbilical arterial blood gas potential of hydrogen<7.0, OR 30 minutes base excess≤-12 mmol/L, OR need for ventilation 5 minutes after birth.
3. All infants must have signs of encephalopathy (such as convulsion, coma, dystonia, abnormal primitive reflex and irregular respiration) within 6 hours of age or continued abnormal EEG for more than 24h.

Exclusion Criteria:

1. Does not meet the inclusion criteria
2. Suffer from other serious organic disease or congenital, hereditary metabolic diseases
3. Intracranial active infection, or neuromuscular damage outside central nervous system
4. potential of hydrogen / electrolyte disorders without improvement or stability
5. Coagulation disorders associated with bleeding tendency
6. Immune function is not perfect
7. Patients or his guardian refuse consent.
8. Patients or his guardian don't accept the follow-up schedule.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal Behavioral Neurological Assessment | 14days after birth
number of adverse events | 7days after cell or factor injection
  adverse events like fever、infection、seizures、hemorrhage coursed by interventions
Neonatal Behavioral Neurological Assessment | 28days after birth

SECONDARY OUTCOMES:
Bayley score | 12 months after birth
  Gross motor function measure assessment for children diagnosed cerebral palsy
Bayley score | 18 months after birth
  Gross motor function measure assessment for children diagnosed cerebral palsy
Peabody development measure scale | 12 months after birth
  Gross motor function measure assessment for children diagnosed cerebral palsy
Peabody development measure scale | 18 months after birth
  Gross motor function measure assessment for children diagnosed cerebral palsy
Number of death | 1 years after birth
Number of participants with treatment-related central nervous tumor as assessed by Magnetic Resonance Imaging or CT | 5 years after birth

CONTACTS AND LOCATIONS:
Overall Officials: Zuo Luan, MD, Study Chair — Navy General Hosiptal
Locations (2):
- China (2):
  - Navy General Hospital, Beijing, Beijing Municipality
  - Navy General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luan Z, Liu W, Qu S, Du K, He S, Wang Z, Yang Y, Wang C, Gong X. Effects of neural progenitor cell transplantation in children with severe cerebral palsy. Cell Transplant. 2012;21 Suppl 1:S91-8. doi: 10.3727/096368912X633806. PMID 22507684
- [Derived] Bruschettini M, Romantsik O, Moreira A, Ley D, Thebaud B. Stem cell-based interventions for the prevention of morbidity and mortality following hypoxic-ischaemic encephalopathy in newborn infants. Cochrane Database Syst Rev. 2020 Aug 19;8(8):CD013202. doi: 10.1002/14651858.CD013202.pub2. PMID 32813884